CLINICAL TRIAL: NCT01091896
Title: Adjuvant Intravitreal Bevacizumab in Pars Plana Vitrectomy for Vitreous Hemorrhage Secondary to Diabetic Retinopathy
Brief Title: Adjuvant Intravitreal Bevacizumab in Pars Plana Vitrectomy for Vitreous Hemorrhage
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Hospital das Clínicas de Ribeirão Preto - University of São Paulo, USP
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IBEViH; IBEViH
Record Dates: First submitted 2010-03-23; First posted 2010-03-24 (Estimated); Last update posted 2010-03-24 (Estimated); Status verified 2010-03

CONDITIONS: Vitreous Hemorrhage Secondary to PDR
Keywords: bevacizumab; vitreous hemorrhage; diabetes mellitus
MeSH Terms: conditions — Vitreous Hemorrhage; Diabetes Mellitus | interventions — Bevacizumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 - no bevacizumab (No Intervention): Patients will not receive bevacizumab before nor during vitrectomy
- 2- bevacizumab before vitrectomy (Experimental): Patients will receive intravitreal injection of 1.25 mg of bevacizumab (0.05 ml) 7 days before vitrectomy
  Interventions: Drug: Bevacizumab
- 3- bevacizumab after vitrectomy (Experimental): Patients will receive intravitreal injection of 1.25 mg of bevacizumab (0.05 ml) at the end of vitrectomy
  Interventions: Drug: bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — 1.25 mg of bevacizumab (0.05 ml) 7 days before vitrectomy
  Arms: 2- bevacizumab before vitrectomy
Drug: bevacizumab — 1.25 mg of bevacizumab (0.05 ml) at the end of vitrectomy
  Arms: 3- bevacizumab after vitrectomy

SUMMARY:
The purpose of this study is to determine the effect of pre and intra-operative bevacizumab injection on postoperative vitreous hemorrhage after diabetic vitrectomy in comparison to vitrectomy without bevacizumab injection.

DETAILED DESCRIPTION:
Postoperative vitreous hemorrhage is a common complication after vitrectomy for proliferative diabetic retinopathy. Bevacizumab (Avastin) is a potent inhibitor of angiogenesis and has been shown to decrease retinal and iris neovascularization in proliferative diabetic retinopathy. We believe that preoperative bevacizumab injection could reduce postoperative vitreous hemorrhage by decreasing the amount of abnormal vessels and intraoperative injection could also reduce postoperative vitreous hemorrhage by inhibiting the vessel formation after surgery

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing first vitrectomy for vitreous hemorrhage secondary to proliferative diabetic retinopathy

Exclusion Criteria:

* follow-up period of less than 3 months
* not first vitrectomy
* abnormal blood coagulation
* uncontrolled hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-09 (Estimated); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
Recurrent vitreous hemorrhage incidence after vitrectomy | 3 months

SECONDARY OUTCOMES:
Visual outcome | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Almeida, MD, Principal Investigator — University of Sao Paulo
Locations (1):
- Hospital das Clínicas de Ribeirão Preto - University of São Paulo, Ribeirão Preto, São Paulo, Brazil

REFERENCES:
- [Background] Tonello M, Costa RA, Almeida FP, Barbosa JC, Scott IU, Jorge R. Panretinal photocoagulation versus PRP plus intravitreal bevacizumab for high-risk proliferative diabetic retinopathy (IBeHi study). Acta Ophthalmol. 2008 Jun;86(4):385-9. doi: 10.1111/j.1600-0420.2007.01056.x. Epub 2007 Nov 7. PMID 17995982
- [Derived] Dervenis P, Dervenis N, Smith JM, Steel DH. Anti-vascular endothelial growth factors in combination with vitrectomy for complications of proliferative diabetic retinopathy. Cochrane Database Syst Rev. 2023 May 31;5(5):CD008214. doi: 10.1002/14651858.CD008214.pub4. PMID 37260074